CLINICAL TRIAL: NCT01980550
Title: Association of Functional COMT Val108/Met Polymorphism With Smoking Cessation in Nicotine Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Dependence, China (Other)
Collaborators: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: Hongqiang-2010
Record Dates: First submitted 2011-04-13; First posted 2013-11-11 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- sublingual nicotine，placebo (Experimental): sublingual nicotine：one or two tablets per hour, up to a maximum of 20 tablets per day Subjects were advised to use the full treatment dose for 4 weeks
  Interventions: Drug: sublingual nicotine

INTERVENTIONS:
Drug: sublingual nicotine — The nicotine sublingual tablet is Smokers were recommended to use one or two tablets per hour, up to a maximum of 20 tablets per day. Subjects were advised to use the full treatment dose for 4 weeks. After this time-point, treatment could be tapered off up to the 8-week visit. During the next 4-week follow-up phase, no further medication was dispensed. Staff, who dispensed medications, were not involved in treating the subjects. During each patient visit, the importance of adequate dosing with study medication was emphasized. The medication was free of charge. In addition, all participants received six sessions of standardized behavioral group counseling focusing on self-monitoring and behavioral modification approaches.
  Other Names: nicotine sublingual tablet

SUMMARY:
Nicotine replacement treatment (NRT) can be efficacious for smoking cessation, but used by only a minority of smokers in China. Pharmacogenetic matching may improve treatment outcomes for NRT in subgroups of smokers. The investigators evaluated the efficacy and safety of sublingual nicotine tablets (SNT) for smoking cessation and the association of catechol-O-methyltransferase (COMT) genotype with efficacy in this smoking cessation trial among Chinese smokers.

DETAILED DESCRIPTION:
All subjects provided written informed consent after a full explanation of the protocol design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects motivated to stop smoking and Han Chinese
* aged 20-70 years who lived in the Haidian District of Beijing
* smoke ≥10 cigarettes/day
* have smoked for ≥3 years
* carbon monoxide (CO) level ≥10 p.p.m. in exhaled air

Exclusion Criteria:

* a history of "Diagnostic and Statistical Manual of Mental Disorders-fourth Edition" (DSM-IV) psychiatric disorder
* alcohol abuse and other drug abuse
* with pathological changes in the floor of their mouth
* cardiovascular disease
* taking psychotropic medications
* using other forms of tobacco or any other NRT products during the last 6 months
* pregnant or breast-feeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-03; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Changes in the exhaled carbon monoxide (CO) level during the 12-week study | The first was 1 day before quit day (baseline), followed by visits after 1, 2, 4, 6 and 8 weeks at the end of treatment (EOT), with a final follow-up visit at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: xiang y zhang, professor, Principal Investigator — VA Medical Center，USA